CLINICAL TRIAL: NCT07055009
Title: Multi-centred Clinico-genetic Study of Actinic Prurigo in Thailand
Status: Recruiting | Type: Observational
Sponsor: Chulalongkorn University (Other)
Collaborators: Health Systems Research Institute,Thailand (Other Government)
Responsible Party: Sponsor
Other Study IDs: CU41/2566
Record Dates: First submitted 2025-06-04; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-05

CONDITIONS: Actinic Prurigo
Keywords: Actinic prurigo; subtype actinic prurigo; HLA typing; genetic
MeSH Terms: conditions — Actinic Prurigo

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case
  Interventions: Diagnostic Test: Targeted long-read HLA sequencing; Other: RNA extraction; Other: Full Skin examination
- Control
  Interventions: Diagnostic Test: Targeted long-read HLA sequencing; Other: RNA extraction

INTERVENTIONS:
Diagnostic Test: Targeted long-read HLA sequencing — Genetic study
  Other Names: Short-read whole genome sequencing
Other: RNA extraction — Nanostring technology, Seattle
Other: Full Skin examination — Skin and mucosa examination
  Groups: Case

SUMMARY:
This research project investigates the clinical and genetic associations of Actinic Prurigo (AP) in the Thai population. As a rare chronic photodermatosis, AP has been observed to occur more frequently in individuals with certain genetic predispositions, particularly specific Human Leukocyte Antigen (HLA) types. Previous studies have suggested variations in clinical presentation and HLA allele distributions between Asian and Western populations.

The primary aim is to explore the relationship between clinical manifestations of AP and genetic profiles, including HLA typing, among Thai individuals. Additionally, the study seeks to examine whether different HLA types are associated with varying responses to treatment.

The study design is a cross-sectional comparative study, involving both AP patients and age-matched healthy controls. Given the rarity of the condition, patient recruitment will be conducted across four collaborating institutions:

King Chulalongkorn Memorial Hospital Siriraj Hospital Institute of Dermatology

ELIGIBILITY:
Inclusion Criteria:

* Thai ethnicity
* Diagnosed with Actinic Prurigo (AP) according to the diagnostic criteria defined for this study
* Mentally competent, able to communicate, and able to read Thai.
* Participants receiving Thalidomide treatment must use two simultaneous methods of contraception, starting at least 4 weeks prior to initiating the medication and continuing throughout the treatment period and for at least 4 weeks after discontinuation.

Exclusion Criteria:

* History and physical examination findings suggestive of other photodermatoses such as Lupus erythematosus, Porphyria, or Polymorphous Light Eruption, among others.
* Elevated Epstein-Barr Virus (EBV) viral load detected in blood testing (EBV viral load will be tested in all participants).
* Low Minimal Erythema Dose (MED) to UVB radiation as the only abnormal finding.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Actinic Prurigo (AP)
Sampling Method: Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Targeted long-read HLA sequencing | through study completion, an average of 1 year
  Correlation between the occurrence of Actinic Prurigo (AP), its clinical manifestations, and genetic factors-including HLA types-in individuals of Thai ancestry.

SECONDARY OUTCOMES:
Short-read whole genome sequencing (WGS) | through study completion, an average of 1 year
  Correlation between the occurrence of Actinic Prurigo (AP), its clinical manifestations, and genetic factors-including short-read whole genome sequencing (WGS)-in individuals of Thai ancestry.
Immunology study | through study completion, an average of 1 year
  Correlation between the occurrence of Actinic Prurigo (AP), its clinical manifestations, and immunological factors in individuals of Thai ancestry, measured by RNA extraction and gene expression analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No